CLINICAL TRIAL: NCT00308308
Title: A Prospective, Multi-Center, Open-Label, Randomized, Controlled Clinical Trial Comparing the Efficacy and Safety in Subjects With Type 1 Diabetes Receiving Subcutaneous Basal Insulin and Prandial Inhalation of Technosphere/Insulin Versus Subcutaneous Basal and Prandial Insulin Over a 52-Week Treatment Period and a 4-Week Follow Up
Brief Title: Efficacy & Safety of Inhaled Insulin in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-009
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes, Type I
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (2):
- 1 (Experimental): Technosphere Insulin
  Interventions: Drug: Technosphere Insulin
- 2 (Active Comparator): Rapid-acting analogue insulin plus basal insulin glargine
  Interventions: Drug: Active comparator

INTERVENTIONS:
Drug: Technosphere Insulin — Inhalation, 15U/30U
  Arms: 1
Drug: Active comparator — sc injectable insulin
  Arms: 2

SUMMARY:
To determine the safety and efficacy of inhaled insulin in the treatment of type 1 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least 1 year
* Nonsmokers for prior 6 months
* BMI less than or equal to 35kg/m2
* HbA1c > or = 7% and < or = 11%
* Serum creatinine < or = 1.8 mg/dL in female subjects and < or = 2.0 mg/dL in male subjects
* FEV1 > or = 70% of predicted, DLco > or = 70% , TLC > or = 80% predicted
* Maintenance of a treatment regimen of insulin less than or equal to 1.4 iu/kg/day
* Urine cotinine < or = 100 ng/mL

Exclusion Criteria:

* History of chronic obstructive pulmonary disease, asthma, any other clinically significant pulmonary disease confirmed by documented history, pulmonary function testing or radiologic findings
* Evidence of severe complications of diabetes
* Aminotransferase and/or alanine aminotransferase > than 3 times the upper limit of normal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (129):
- United States (61):
  - Coastal Clinical Research Inc, Mobile, Alabama
  - Radiant Research (Phoenix), Chandler, Arizona
  - International Clinical Research Network, Chula Vista, California
  - Family Medical Center, Foothill Ranch, California
  - Diabetes/Lipid Management and Research Center, Huntington Beach, California
  - South Bay Clinical Research, Inglewood, California
  - Radiant Research, San Diego, California
  - Coastal Biomedical Research Inc, Santa Monica, California
  - Diabetes Research Center, Tustin, California
  - International Research Associates LLC, Miami, Florida
  - Laureate Clinical Research Group, Atlanta, Georgia
  - Atlanta Pharmaceutical Research Center, Dunwoody, Georgia
  - North Atlanta Endocrinology & Diabetes PC, Lawrenceville, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - John H Stoger Jr Hospital of Cook County, Chicago, Illinois
  - Clintell Inc, Skokie, Illinois
  - Medical Research of Louisiana, Metairie, Louisiana
  - Oschner Clinic Foundation, New Orleans, Louisiana
  - James A Dicke MDPA, Towson, Maryland
  - Wayne State University, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Michigan Institute of Medicine, Livonia, Michigan
  - KMED Research, Saint Clair Shores, Michigan
  - Radiant Research Inc (Minneapolis), Edina, Minnesota
  - International Diabetes Center, Minneapolis, Minnesota
  - Center for Urologic Clinical Trials University of Minnesota, Minneapolis, Minnesota
  - Amin Radparvar's Private Practice, City of Saint Peters, Missouri
  - Healthcare Research, Florissant, Missouri
  - MedEx Healthcare Research Inc(009), St Louis, Missouri
  - Billings Clinic Research Division, Billings, Montana
  - Creighton Diabetes Center, Omaha, Nebraska
  - University of New Mexico HCS, Albuquerque, New Mexico
  - Winthrop University Hospital, Mineola, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - University of Physicians Group Endocrine Division, Staten Island, New York
  - Endocrine Research - Physician's East PA, Greenville, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Health Partners - Center of Clinical Research, Dayton, Ohio
  - Portland Diabetes & Endocrinology Center, Portland, Oregon
  - Legacy Clinical Research, Portland, Oregon
  - Covance CRU Inc., Portland, Oregon
  - Pennsylvania Research Institute, Bensalem, Pennsylvania
  - Southeastern Research Associates Inc, Williamston, South Carolina
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - The Endocrine Clinic, Memphis, Tennessee
  - Israel Hartman MD, Arlington, Texas
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - Radiant Research Dallas-North, Dallas, Texas
  - Baylor Endocrine Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Spuhler Medical Associates, Friendswood, Texas
  - Quality Assurance Research Center (900), San Antonio, Texas
  - Diabetes & Glandular Disease Research Assoc PA, San Antonio, Texas
  - SAM Clinical Research Center, San Antonio, Texas
  - Edward Bali MD PA, Seguin, Texas
  - Radiant Research Salt Lake City, Salt Lake City, Utah
  - Salt Lake Research, Salt Lake City, Utah
  - Sentara Medical Group, Virginia Beach, Virginia
  - Larry D Stonesifer MD Inc PS, Federal Way, Washington
  - Cedar Research, Tacoma, Washington
  - Liberty Research Center, Tacoma, Washington
- Argentina (8):
  - Hospital Interzonal de Agudos Pedro Fiorito, Avellaneda, Buenos Aires
  - Centro Endocrinologic Tiempo, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Durand /Buenos Aires, Buenos Aires
  - Hospital Gral De Agudos Dr. Teodoro Alvarez, Buenos Aires
  - Cons Asoc de Endocrinologia, Buenos Aires
  - Centro Medico Dra De Salvo, Buenos Aires
  - CIMeL, Buenos Aires
- Brazil (11):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - CPClin-Centro de Pesquisas Clinicas, São Paulo, São Paulo
  - Universidade Estabual de Maringa, Maringa Parana
  - Nucleo de Medicina Integrada, Mogi das Cruzes
  - Instituto Estadual De Diabetes e Endocrinologia Luis Capriglione, Rio de Janeiro
  - Ccbr Brasil Centro de Analises e Pesquisas Clinicas Ltda, Rio de Janeiro
  - Hospital Guilherme Alvaro, Santos
  - Centro de Diabetes/UNIFESP-EPM, São Paulo
  - Blumenau Servicos Medicos S/C Ltda, São Paulo
  - Instituto de Pesquisa Clinica e Medicina Avancada, São Paulo
- Canada (4):
  - Lifestyle Metabolism Center, Oakville, Ontario
  - Lifestyle Metabolism Center, Thornhill, Ontario
  - Lifestyle Metabolism Center, Toronto, Ontario
  - Windsor Professional Research, Windsor, Ontario
- Chile (6):
  - Hospital del Salvador, Santiago, Santiago Metropolitan
  - Hospital San Jose, Santiago
  - Hospital Clinico Pontificia Universidad (009)Catolica de Chile, Santiago
  - Hospital Padre Alberto Hurtado, Santiago
  - Hospital San Borja ArriaranUniversidad de Chile, Santiago
  - Instituto de Informacion de Tramiento y Educacion en Salud, Santiago
- Mexico (5):
  - Instituto Mexicano de Investigacion, Mexico City, Durango
  - Hospital Santa Engracia-CIMA, Garza García
  - Centro de Estudios en Diabetes, Mexico City
  - Hospital General de Mexico Servicio EndocrinologiaJefe Del Servicio, Mexico City
  - Hospital OCA-MIRC (009), Monterrey
- Poland (7):
  - NZOZ Specjalistyczny Osrodek Internistyczno - Diabetologiczny, Bialystok, POL
  - Katedra I Klinika Chorob Metabolicznych Collegium Medicum Uniwersytety Jagiellonskiego, Krakow, POL
  - Instytut Centrum Zdrowia (009) Matki Polki, Lodz, POL
  - Szpital Kolejowy im Dr w Roeflera(009) Oddzial Gastorenterologii, Pruszków, POL
  - Oddzial Chorob Wewnetrznych (009 Endokrynologii I Diabetologii Szpitala Wojewodzkiego, Bialystok
  - Oddzial Kliniczny Diabetologii (009) Kliniczny nr 1 im Norberta Barlickiego Uniwersytety Meycznego, Lodz
  - NZOZ Diabetologiczna Poradnia Specjalistyczna, Warsaw
- Russia (17):
  - NHI Kemerovo Regional Clinical Hospital, Kemerovo, RUS
  - NI Principal Military Clinical Hospital n a academician N.N. Burdenko of the Ministry of Defense, Moscow, RUS
  - NEI HPE Moscow State University of Medicine and Dentistry of FAHSD City Clinical Hospital #70, Moscow, RUS
  - Moscow City Clinical Hospital # 13, Moscow, RUS
  - SEI HPE Moscow Medical Academy IM Sechenov of Roszdrav Clinic of Endocrinology, Moscow, RUS
  - SI Internal Affairs of Moscow- Clinical Hospital, Moscow, RUS
  - RAAMS Endocrinology and Diabetology Department, Moscow, RUS
  - SIH of Moscow City Clinical Hopsital #81Endocrinology and Diabetology, Moscow, RUS
  - St Petersburg NHI City Polytclinic #77 City Diabetological Center #4, Saint Petersburg, RUS
  - Central Medical Sanitary Unit #122, Saint Petersburg, RUS
  - St Petersburg NHI Municipal Multi-Speciality Hospital # 2, Saint Petersburg, RUS
  - Pavlov State Medical Univ of St Petersburg, Saint Petersburg, RUS
  - MHI Clinical Hospital for Emergency Care na NV Soloviev, Yaroslavl, RUS
  - MCHI Medical Sanitary Unit of Novo-Yaroslavsky Oil Refining Plant, Yaroslavl, RUS
  - NHI Yaroslavl Regional Clinical Hospital, Yaroslavl, RUS
  - City Clinical Hospital # 61, Moscow
  - Russian Scientific Center of Restoration Medicine & Balneology, Moscow
- Spain (5):
  - Complejo Hospitalario Nuestra Senora de Valme, Seville, Andalusia
  - Hospital del Mar, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Complejo Hospitalario Virgen del Rocio, Seville
  - Hospital Virgen Macarena (policlinico) 2ª planta Servicio de Endocrinologia y Nutricion, Seville
- United Kingdom (5):
  - Birchwood Surgery, Letchworth Garden City, Herts
  - Lister Hospital, Stevenage, Herts
  - Sandwell General Hospital, Lyndon, West Bromwich
  - Guy's & St Thomas Hospital, London
  - Yaxley Group Practice, Peterborough

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient enrolled Feb, 2006 Multi-national trial conducted in US, Canada, Mexico, Brazil, Argentina, Chile, Spain, UK, Poland, Russia
Pre-assignment Details: 3 week Screening Period prior to randomization - 1420 Screened / 598 Eligible of which 589 were randomized - 822 screen failures 24 Subjects randomized but never dosed
Groups:
- TI + Insulin Glargine: TI + Insulin glargine
- Insulin Aspart + Insulin Glargine: Comparator
Period: Overall Study
Arm/Group | TI + Insulin Glargine | Insulin Aspart + Insulin Glargine
Started | 301 | 288
Completed | 198 | 220
Not Completed | 103 | 68
Not completed — Adverse Event | 17 | 2
Not completed — Lost to Follow-up | 5 | 5
Not completed — Physician Decision | 15 | 7
Not completed — Protocol Violation | 3 | 14
Not completed — Withdrawal by Subject | 47 | 19
Not completed — Various | 7 | 5
Not completed — Randomized but not dosed | 8 | 16
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population (589 were randomized - 24 Subjects randomized but never dosed)
Groups:
- Total: Total of all reporting groups
Arm/Group | TI + Insulin Glargine | Insulin Aspart + Insulin Glargine | Total
Number analyzed (Participants) | 293 | 272 | 565
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (13.06) | 38.1 (13.18) | 38 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 132 | 271
  Male | 154 | 140 | 294
HbA1c [Mean (Standard Deviation); unit: percent] — Glycosylated Hemoglobin
  percent | 8.4 (0.95) | 8.5 (0.97) | 8.5 (0.96)
Weight [Mean (Standard Deviation); unit: kilogram] — Weight in kilograms
  kilogram | 76.7 (15.64) | 76.8 (14.95) | 76.7 (15.3)

OUTCOME MEASURES:

1. Primary Outcome: Compare the Mean Change From Baseline to Week 52 in HbA1c
Time Frame: Baseline to Week 52
Population: Intention to treat (ITT) with Last Observation Carried Forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | TI + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 277 | 262
Percentage | -0.13 (0.058) | -0.37 (0.059)
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs Insulin Aspart + Insulin Glargine; Test type: Non-Inferiority or Equivalence — Sample size was set to meet regulatory requirement of 250 subjects per arm with 52-week data, resulting in > 90% power for a non-inferiority test of the difference in 12-month change of HbA1c scores between treatment groups with non-inferiority margin of 0.4%, standard deviation of 1.2 and 1-sided alpha of 0.025. Allowing for a 15% dropout rate, 589 subjects were randomized; ANCOVA; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [0.08 to 0.40], Standard Error of Mean 0.082

2. Secondary Outcome: Change From Baseline in Weight to Week 52
Description: Change from baseline in weight at Week 52
Time Frame: Baseline to Week 52
Population: participants in ITT population with available data
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | TI + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 186 | 206
kilogram | -0.5 (0.32) | 1.4 (0.30)
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs Insulin Aspart + Insulin Glargine; ANCOVA model with terms of pooled site and treatment as fixed effects and baseline weight as covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -1.8, 95% CI [-2.7 to -1.0], Standard Error of Mean 0.42

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose to Week 52
Description: Change from baseline in fasting plasma glucose at Week 52
Time Frame: Baseline to Week 52
Population: participants in ITT population with available data
Measure: Least Squares Mean (Standard Error); unit: mg/dl
Arm/Group | TI + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 178 | 195
mg/dl | -46.5 (5.61) | -25.7 (5.23)
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs Insulin Aspart + Insulin Glargine; Test type: Superiority or Other; p = 0.0052, ANCOVA; Mean Difference (Net) = -20.9, 95% CI 2-sided [-35.4 to -6.3], Standard Error of Mean 7.41

4. Secondary Outcome: Number of Subjects Achieving Week 52 HbA1c Levels Less Than or Equal to 7.0%
Description: Number of subjects achieving week 52 HbA1c levels less than or equal to 7.0%
Time Frame: Baseline to Week 52
Population: participants in ITT population with available data
Measure: Number; unit: Participants
Arm/Group | TI + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 202 | 219
Participants | 33 | 35
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs Insulin Aspart + Insulin Glargine; logistic regression analysis with the terms of treatment and baseline HbA1c in the model; Test type: Superiority or Other; p = 0.8311, Regression, Logistic; Odds Ratio (OR) = 0.941, 95% CI 2-sided [0.536 to 1.652]

5. Secondary Outcome: Incidence of Total Hypoglycemia
Description: Defined as hypoglycemic symptoms that are relieved with carbohydrate intake or blood glucose measurement <= 63 mg/dL, regardless of symptoms.
Time Frame: Baseline to Week 52
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | TI + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 293 | 272
percentage of participants | 85.67 | 92.28
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs Insulin Aspart + Insulin Glargine; Test type: Superiority or Other; p = 0.0124, Regression, Logistic; Odds Ratio (OR) = 0.488, 95% CI 2-sided [0.278 to 0.856] — Model: Treatment + Site

6. Secondary Outcome: Incidence of Severe Hypoglycemia
Description: Severe hypoglycemia occurs when all 3 of the following occur simultaneously:
  * Subject requires the assistance of another person;
  * Subject exhibits at least 1 cognitive neurological symptom (memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, seizure, loss of consciousness);
  * Measured BG is ≤ 49 mg/dL (2.7 mmol/L), or, in the absence of a BG measurement, clinical symptoms are reversed by oral carbohydrates, sc glucagon or intravenous glucose administration; OR,
  * Measured BG is ≤ 36 mg/dL (2.0 mmol/L) with or without symptoms.
Time Frame: Baseline to Week 52
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | TI + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 293 | 272
percentage of participants | 32.08 | 36.40
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs Insulin Aspart + Insulin Glargine; Test type: Superiority or Other; p = 0.2786, Regression, Logistic; Odds Ratio (OR) = 0.825, 95% CI 2-sided [0.582 to 1.169] — Model: Treatment + Site

7. Secondary Outcome: Total Hypoglycemia Event Rate
Description: Number of Hypoglycemic Events/Total Subject Exposure Time (in months)
Time Frame: Baseline to Week 52
Population: Safety Population
Measure: Number; unit: Number of events/subject-month
Arm/Group | TI + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 293 | 272
Number of events/subject-month | 1.81 | 1.86
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs Insulin Aspart + Insulin Glargine; Test type: Superiority or Other; p = 0.1193, Generalized Estimation Equation; * Based on Poisson distribution * Model: Treatment + Time Period

8. Secondary Outcome: Severe Hypoglycemia Event Rate
Description: Number of Severe Hypoglycemic Events/Total Subject Exposure Time (in months)
Time Frame: Baseline to Week 52
Population: Safety Population
Measure: Number; unit: Number of events/subject-month
Arm/Group | TI + Insulin Glargine | Insulin Aspart + Insulin Glargine
Number analyzed (Participants) | 293 | 272
Number of events/subject-month | 0.08 | 0.10
Statistical Analysis 1: Comparison: TI + Insulin Glargine vs Insulin Aspart + Insulin Glargine; Test type: Superiority or Other; p = 0.2131, Generalized Estimating Equation; * Based on Poisson distribution * Model: Treatment + Time Period

ADVERSE EVENTS:
Time Frame: From first dose to 30 days after last dose
Description: Safety population is the at risk population
Arm/Group | TI + Insulin Glargine | Insulin Aspart + Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 52/293 | 47/272
Other Adverse Events (participants affected / at risk) | 265/293 | 257/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TI + Insulin Glargine (N=293) | Insulin Aspart + Insulin Glargine (N=272)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hepatocellular damage (Hepatobiliary disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 30 | 34
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 2 | 4
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 3 | 0
Localised infection (Infections and infestations) | 0 | 1
Loss of consciousness (Nervous system disorders) | 8 | 7
Metabolic syndrome (Metabolism and nutrition disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TI + Insulin Glargine (N=293) | Insulin Aspart + Insulin Glargine (N=272)
Cough (Respiratory, thoracic and mediastinal disorders) | 98 | 21
Headache (Nervous system disorders) | 16 | 15
Hypoglycaemia (Metabolism and nutrition disorders) | 252 | 252
Influenza (Infections and infestations) | 23 | 19
Nasopharyngitis (Infections and infestations) | 37 | 38
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 6
Pulmonary function test decreased (Investigations) | 16 | 4
Upper respiratory tract infection (Infections and infestations) | 46 | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MannKind has right to 1st joint multicenter publication. After 1st publication PI may publish data only if PI submits proposed publication to MNKD for review 60 days prior to publication date. MNKD may remove any confidential information. If a multicenter publication is not submitted 12 months after conclusion, abandonment, or termination of the Study at all sites, or if MNKD confirms there will be no multicenter Study publication, PI may publish the Study results subject to MNKD rights herein.